CLINICAL TRIAL: NCT02953717
Title: A Prospective Randomized Study to Compare Cognitive Outcome After Stereotactic Radiosurgery or Whole Brain Radiation Therapy in Patients With 11-20 Brain Metastases
Brief Title: Cognitive Outcome After SRS or WBRT in Patients With Multiple Brain Metastases (CAR-Study B)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Tilburg University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 842003006; NTR5463 (Registry Identifier: Netherlands Trail Register)
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-05

CONDITIONS: Neoplasm Metastasis
Keywords: Brain metastases; Cognition; Radiosurgery; Gamma Knife Radiosurgery; Stereotactic radiosurgery; Whole Brain Radiation Therapy; Quality of Life; Fatigue; Anxiety; Depression
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms; Fatigue; Anxiety Disorders; Depression | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stereotactic radiosurgery (SRS) (Active Comparator): Gamma Knife radiosurgery
  Interventions: Radiation: Gamma Knife radiosurgery
- Whole Brain Radiation Therapy (WBRT) (Active Comparator): Whole Brain Radiation Therapy
  Interventions: Radiation: Whole Brain Radiation Therapy

INTERVENTIONS:
Radiation: Gamma Knife radiosurgery — GKRS is performed with a Leksell Gamma Knife® Icon, Elekta Instruments, AB. Depending upon the volume, a dose of 18-25 Gy will be prescribed with 99-100% coverage of the target.
  Arms: Stereotactic radiosurgery (SRS)
Radiation: Whole Brain Radiation Therapy — Patients in the WBRT group will receive 4 Gy x 5 fractions (total of 20 Gy) in one week, which is a commonly utilized treatment schedule according to Dutch guidelines.
  Arms: Whole Brain Radiation Therapy (WBRT)

SUMMARY:
Whole Brain Radiation Therapy (WBRT) has long been the mainstay of treatment for patients with multiple brain metastases (BM). Meanwhile, Gamma Knife radiosurgery (GKRS) has been increasingly employed in the management of multiple BM to spare healthy tissue. Hence, GKRS is expected to cause fewer cognitive side effects than WBRT. Treatment of multiple BM without cognitive side effects is becoming more important, as more patients live longer due to better systemic treatment options. There are no published randomized trials yet directly comparing GKRS to WBRT in patients with multiple BM, including objective neuropsychological testing.

CAR-Study B is a prospective randomized trial comparing cognitive outcome after GKRS or WBRT in eligible patients with 11-20 BM.

DETAILED DESCRIPTION:
CAR-Study B is a prospective randomized trial comparing cognitive outcome after GKRS or WBRT in eligible patients with 11-20 BM on a triple dose gadolinium-enhanced MRI-scan. Neuropsychological assessment will be performed at baseline and at 3, 6, 9, 12 and 15 months after treatment. Follow-up assessments will be combined with 3-monthly MRI-scans.

Patients will be randomized to either GKRS or WBRT. Groups will be balanced at baseline (prior to radiotherapy), taking into account several (stratification) factors that may influence cognitive functioning over time, such as: total tumor volume in the brain, systemic treatment, KPS, age, histology, and baseline HVLT-R total recall score.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant cancer
* 11-20 newly diagnosed brain metastases on a triple dose gadolinium-enhanced MRI-scan
* Maximum total tumor volume ≤ 30 cm3
* Lesion ≥ 3 mm from the optic apparatus
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) ≥ 70
* Anticipated survival > 3 months

Exclusion Criteria:

* No prior histologic confirmation of malignancy
* Primary brain tumor
* A second active primary tumor
* Small cell lung cancer (SCLC)
* Lymphoma
* Leukemia
* Meningeal disease
* Progressive, symptomatic systemic disease without further treatment options
* Prior brain radiation
* Prior surgical resection of BM
* Cardiovascular accident (CVA) < 2 years ago
* Additional history of a significant neurological or psychiatric disorder
* Contra indications to MRI or gadolinium contrast
* Underlying medical condition precluding adequate follow-up
* Participation in a concurrent study in which neuropsychological testing and/or health-related QOL assessments are involved
* Lack of basic proficiency in Dutch
* IQ below 85
* Severe aphasia
* Paralysis grade 0-3 according to MRC scale (Medical Research Council)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-02; Primary Completion 2023-07 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline at 3 months | 3 months
  Cognitive decline is defined as a significant decline (5 point decrease from baseline based on the Reliable Change Index (RCI) with correction for practice effects) in HVLT-R Total Recall score (verbal learning and memory test) after treatment with either GKRS or WBRT in patients with 11-20 brain metastases at time of treatment initiation.

SECONDARY OUTCOMES:
Verbal memory | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Verbal memory is measured with the Hopkins Verbal Learning Test-Revised (HVLT-R)
Cognitive flexibility | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Cognitive flexibility is measured with the Controlled Oral Word Association (COWA)
Word Fluency | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Word Fluency is measured with the Controlled Oral Word Association (COWA)
Working memory | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Working memory is measured with the Wechsler Adult Intelligence Scale - Digit Span
Processing speed | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Processing speed is measured with the Wechsler Adult Intelligence Scale - Digit Symbol
Motor dexterity | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Motor dexterity is measured with the Grooved Pegboard (GP)
Health Related Quality Of Life (HRQOL) | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is used to measure HRQOL.
Fatigue | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Fatigue is measured with the Multidimensional Fatigue Inventory (MFI).
Depression and anxiety | Baseline and 3, 6, 9, 12 and 15 months post GKRS/WBRT
  Depression and anxiety are measured with the Hospital Anxiety and Depression Scale (HADS).
Median Overall Survival | 12 months after GKRS/WBRT
  Overall survival is defined as the time in months from the start of treatment to the date of death or last contact if alive. Kaplan-Meier methods are used to estimate overall survival.
Local tumor control | 12 months after GKRS/WBRT
  Local brain tumor control of the initial treated lesions is defined as a complete, partial, or stable response, or less than a 25% increase in diameter on contrast-enhanced MRI follow-up and not requiring resection. Any initial treated lesions increased by more than 25% in diameter on contrast-enhanced MRI or required resection will be considered a local failure.
Distant tumor control | 12 months after GKRS/WBRT
  Distant brain tumor control is defined as the absence of any new brain metastases, distinct from the initial treated lesion(s), on follow-up MRI. The appearance of one or more new lesions in the brain by contrast-enhanced follow-up MRI is considered distant failure.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick EJ Hanssens, MD, Principal Investigator — Gamma Knife Center Tilburg, Elisabeth-TweeSteden Hospital, The Netherlands
Locations (1):
- Gamma Knife Center Tilburg, Elisabeth-TweeSteden Hospital, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schimmel WCM, Verhaak E, Hanssens PEJ, Gehring K, Sitskoorn MM. A randomised trial to compare cognitive outcome after gamma knife radiosurgery versus whole brain radiation therapy in patients with multiple brain metastases: research protocol CAR-study B. BMC Cancer. 2018 Feb 21;18(1):218. doi: 10.1186/s12885-018-4106-2. PMID 29466961